CLINICAL TRIAL: NCT04220814
Title: Evaluation of the Impact of Lesions of the Motor and Proprioceptive Brain and Pan-medullary Pathways on Their Clinically and Electrophysiologically Assessed Function in Multiple Sclerosis
Acronym: MS-TRACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC19_9769_MS-TRACTS
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; MRI; pronostic
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental)
  Interventions: Radiation: MRI; Other: Electrophysiology
- Healthy Volunteer (Other)
  Interventions: Radiation: MRI; Other: Electrophysiology

INTERVENTIONS:
Radiation: MRI — MRI protocol is different, a little bit longer than MRI in routine for patients. For healthy volunteer, a specific MRI for this study is done
Other: Electrophysiology — Electrophysiology will be done during routine visits for patients and during inclusion visit to healthy volunteers

SUMMARY:
Multiple Sclerosis (MS) is the most common acquired neurological disease leading to disability, especially ambulatory, in young adults. To date, the correlation between the number or volume of white matter lesions seen on conventional MRI and the degree of disability of patients remains low to moderate. This phenomenon is known as the "clinical-radiological paradox".

In this new project, we hypothesize that an evaluation of the corticospinal pathways including their thoracic medullary portion, as well as taking into account the severity of the lesions using quantitative MRI, will allow the investigators to refine the correlation with ambulatory disability in MS patients. We will complete the evaluation of motor pathways with those of the proprioceptive pathways also strongly involved in ambulation.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is the most common acquired neurological disease leading to disability, especially ambulatory, in young adults. To date, the correlation between the number or volume of white matter lesions seen on conventional MRI and the degree of disability of patients remains low to moderate. This phenomenon is known as the "clinical-radiological paradox".

The impact of the precise localisation of focal MS lesions on certain circuits particularly involved in ambulation, such as pyramidal or proprioceptive beams, has however been little studied in imaging, mainly due to technical limitations. Indeed, such studies require the acquisition of brain and spinal cord MRI images of sufficient spatial resolution to allow the localisation of focal lesions and pathways. Several previous studies have shown encouraging results by separately studying damage to the brain or spinal cord portion of the corticospinal bundle and relating it to disability. To our knowledge, no studies have analysed the lesional involvement of the cortico-spinal bundle or the entire proprioceptive bundle from the motor cortex to the medullary cone in patients with MS.

In a preliminary study, we studied the cerebral spinal cortex and cervical spinal cord bundle using data from the PHRC 2012 EMISEP and obtained encouraging results. In particular, we have shown that the cortico-spinal pathways are very frequently affected by focal lesions in the early years of the disease and that it is already correlated with the functional consequences in patients measured clinically and in electrophysiology.

In this new project, we hypothesize that an evaluation of the corticospinal pathways including their thoracic medullary portion, as well as taking into account the severity of the lesions using quantitative MRI, will allow the investigators to refine the correlation with ambulatory disability in MS patients. We will complete the evaluation of motor pathways with those of the proprioceptive pathways also strongly involved in ambulation.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* More than 18 years old
* relapsing-remitting multiple sclerosis according to Mac Donald criteria (2010)
* EDSS score at the inclusion from 0 to 4
* With at least 1 symptom of pyramidal injury during clinical exam
* Written informed consent
* Affiliated to a Health Care system

Healthy Volunteers:

* More than 18 years old
* Written informed consent
* Affiliated to a Health Care system

Exclusion Criteria:

Patients

* progressive MS ;
* Corticoids during the last 60 days before inclusion ;
* Other neurological disease or Other progressive systemic disease
* adults subject to legal protection or persons deprived of liberty
* Contraindications to MRI
* Contraindications to motor evoked potentials
* Current pregnancy or breast-feeding

Healthy volunteers:

* History of disease affecting central nervous system
* Familial history of MS
* History of medullar injury
* Spinal osteoarthritis which can lead to a spinal hypersignal ;
* adults subject to legal protection or persons deprived of liberty
* Contraindications to MRI
* Contraindications to motor evoked potentials
* Current pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
association ratio between EDSS score and focal injury fraction at inclusion | 24 months
  EDSS score is a specific multiple sclerosis scale, named Expanded Disability Status Scale, from 0 (normal neurological status) to 10 (death kinked to sclerosis). Focal injury fraction is focal injury volume divided by the volume of goal zone and will be assessed by MRI analysis.

SECONDARY OUTCOMES:
Correlation between focal lesion load and changes in Expanded Disability Status Scale (EDSS) | 24 months
  Correlation between focal lesion load and changes in Expanded Disability Status Scale (EDSS) during patients follow up. The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Correlation between the severity of lesions and changes in Expanded Disability Status Scale (EDSS) | 24 months
  Correlation between the severity of lesions and changes in Expanded Disability Status Scale (EDSS) during patients follow up. The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
  The severity of the lesions will be assessed by the volume of the focal lesion load on the motor and sensory pathways, and by the value of the average magnetization transfer ratio (MTR) within the lesions
Differences in central conduction times between patients and healthy volunteers | 1 day
  Significance of the differences in central conduction time values of motor and somaesthetic evoked potentials and in mean MTR values of motor and sensory pathways, between patients and healthy volunteers. Central conduction time values of motor and somaesthetic evoked potentials in healthy subjects and patients as well as on the averages of MTR (magnetic transfer ratio) values of motor and sensory pathways at the encephalic and medullary level, between patients and healthy volunteers
Correlation between focal lesion load and changes in Timed 25-Foot Walk Test (T25W) | 24 months
  Correlation between focal lesion load and changes in Timed 25-Foot Walk Test (T25W) during patients follow up. The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. It is the first component of the MSFC to be administered at each visit. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible. he task is immediately administered again by having the patient walk back the same distance. The score for the T25-FWis the average of the two completed trials.
Correlation between the severity of lesions and changes in Timed 25-Foot Walk Test (T25W) | 24 months
  Correlation between the severity of lesions and changes in Timed 25-Foot Walk Test (T25W) during patients follow up. The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. It is the first component of the MSFC to be administered at each visit. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible. he task is immediately administered again by having the patient walk back the same distance. The score for the T25-FWis the average of the two completed trials.The severity of the lesions will be assessed by the volume of the focal lesion load on the motor and sensory pathways, and by the value of the average magnetization transfer ratio (MTR) within the lesions
Correlation between focal lesion load and changes in Nine Hole Peg Test (9HPT) | 24 months
  Correlation between focal lesion load and changes in Nine Hole Peg Test (9HPT) during patients follow up. The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnose. Scores are based on the time taken to complete the test activity, recorded in seconds
Correlation between the severity of lesions and changes in Nine Hole Peg Test (9HPT) | 24 months
  Correlation between the severity of lesions and changes in Nine Hole Peg Test (9HPT) during patients follow up. The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnose. Scores are based on the time taken to complete the test activity, recorded in seconds. The severity of the lesions will be assessed by the volume of the focal lesion load on the motor and sensory pathways, and by the value of the average magnetization transfer ratio (MTR) within the lesions
Correlation between focal lesion load and changes in walking distance | 24 months
  Correlation between focal lesion load and changes in walking distance using 6-minutes walk test (6MWT) during patients follow up. The score of the test is the distance a patient walks in 6 minutes.
Correlation between the severity of lesions and changes in walking distance | 24 months
  Correlation between the severity of lesions and changes in walking distance using 6-minutes walk test (6MWT) during patients follow up. The score of the test is the distance a patient walks in 6 minutes. The severity of the lesions will be assessed by the volume of the focal lesion load on the motor and sensory pathways, and by the value of the average magnetization transfer ratio (MTR) within the lesions
Correlation between focal lesion load and changes in 12-Item Multiple Sclerosis Walking Scale (MSWS12) score | 24 months
  Correlation between focal lesion load and changes in 12-Item Multiple Sclerosis Walking Scale (MSWS12) during patients follow up. The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a patient-reported outcome that assesses the impact of walking impairment in people with multiple sclerosis. The EQ-5D-3L is a validated, generic, preference-based, health-status measure consisting of five descriptive questions encompassing five domains of HRQoL (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each question is answered based on three response options (1= "no problems", 2= "moderate problems", 3= "severe problems"), with the 243 potential patterns of responses enabling classification of a participant into a distinct health state associated with a specific index score.
Correlation between the severity of lesions and all limbs electrophysiology parameters | 24 months
  Correlation between the severity of lesions and all limbs electrophysiology parameters : Electrophysiology (all 4 limbs) with the central conduction time of motor evoked potentials and the central conduction time of somesthetic evoked potentials. The severity of the lesions will be assessed by the volume of the focal lesion load on the motor and sensory pathways, and by the value of the average magnetization transfer ratio (MTR) within the lesions
Correlation between in focal lesion load of pathways and changes in Expanded Disability Status Scale | 24 months
  The amount of focal lesion load in the motor and proprioceptive pathways will be correlated with the change in Expanded Disability Status Scale (EDSS) score during patients follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Chouteau, Md, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - AP-HM Timone, Marseille
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No